CLINICAL TRIAL: NCT05235009
Title: LEVANTIS-0087A: GAGomes for Multi-Cancer Early Detection in Asymptomatic Adults (LEV87A)
Acronym: LEV87A
Status: Recruiting | Type: Observational
Sponsor: Elypta (Industry)
Responsible Party: Sponsor
Other Study IDs: GR 21-063
Record Dates: First submitted 2022-02-07; First posted 2022-02-10 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer
Keywords: liquid biopsy; multi-cancer early detection; glycosaminoglycans
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biobanked plasma and urine biospecimens, originally collected by the selected biobank(s).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sub-Study 1: Adults >= 18 years old with cancer or imminent cancer diagnosis (cases) versus cancer-free and no imminent cancer diagnosis (controls).
  Sub-Study 1 is intended for the development of 3 free GAGome MCED tests.
  Interventions: Diagnostic Test: Combined free GAGome MCED test
- Sub-Study 2: Adults between 35 - 80 years old asymptomatic for cancer and with no recent history of cancer (> 5 years since curative-intent treatment for cancer).
  Sub-Study 2 is intended for the validation of the combined free GAGome MCED test (primary endpoint) and the plasma and urine free GAGome MCED tests (secondary endpoints).
  Interventions: Diagnostic Test: Combined free GAGome MCED test

INTERVENTIONS:
Diagnostic Test: Combined free GAGome MCED test — The combined free GAGome MCED test aggregates measurements of plasma and urine GAGomes (the exhaustive human glycosaminoglycan profile) into a diagnostic score, the combined free GAGome MCED score. The measurements are performed using MIRAM MCED Kits (Elypta AB) and the scores are computed using Elypta SKY Software (Elypta AB)

SUMMARY:
LEVANTIS-0087A (LEV87A) is a retrospective in vitro diagnostics clinical validation population cohort-based case-control study to validate the diagnostic performance of free GAGome-based tests for multi-cancer early detection (MCED) in adults asymptomatic for cancer and with no recent history of cancer.

DETAILED DESCRIPTION:
Multi-cancer early detection (MCED) could prevent 26% of all cancer-related deaths - an effect larger than averting all deaths from breast cancer alone. However, a societal program to implement MCED requires a practical, noninvasive, and affordable diagnostic modality that is sensitive and specific to all forms of cancers. Liquid biopsies represent front-runner modalities to this end but virtually all of them rely on genomics biomarkers, typically circulating free DNA (cfDNA), which capture <20% of cancers in stage I. In addition, they miss certain cancer types that shed little cfDNA, like brain or genitourinary tumors. Pilot studies show that free glycosaminoglycan profiles in plasma and urine, or free GAGomes, were promising noninvasive biomarkers of cancer metabolism that detected over a third of stage I cancers across 14 types, including brain and genitourinary tumors.

LEVANTIS-0087A (LEV87A) is a retrospective in vitro diagnostics clinical validation population cohort-based case-control study to develop free GAGome-based tests for multi-cancer early detection in adults asymptomatic for cancer and with no recent history of cancer (Sub-Study 1) and to validate their diagnostic performance in the target population (Sub-Study 2).

LEV87A uses retrospectively collected biospecimens from one or more population-based biobanks representative of the target population.

ELIGIBILITY:
Sub-Study 1

Inclusion Criteria

* Case Arm:

  * At the baseline visit, >18 years old, any gender
  * At the baseline visit, available biospecimens for both EDTA-plasma and urine
  * Diagnosis of cancer before or at the baseline visit or diagnosis of cancer after the baseline visit
  * If a diagnosis of cancer before or at the baseline visit, then no antineoplastic treatment between the date of diagnosis and the baseline visit
* Control Arm:

  * At the baseline visit, >18 years old, any gender
  * Not receiving treatment for or under surveillance for cancer at the baseline visit
  * No indications of being monitored for or under consideration for suspected cancer at the baseline visit
  * No diagnosis of cancer before or on the baseline visit or if any previous diagnosis of cancer, then cancer must have been curatively treated ≥ 5 years before the baseline visit
  * No diagnosis of cancer within at least 365 days after the baseline visit
  * At the baseline visit, available biospecimens for both EDTA-plasma and urine
* Exploratory Arm:

  * Same as Control Arm and type 2 diabetes or hypertension or BMI > 30 at the baseline visit

Exclusion Criteria

* Case Arm:

  * No available data for diagnosis of cancer starting 90 days before the baseline visit and up to 365 days after the baseline visit
  * A subject with only a self-reported diagnosis of cancer (either in the 90 days before or in the 365 days after the baseline visit), and absence of a histopathological or clinically indicated diagnosis of cancer, according to biobank database(s), or through linkage with cancer registry(ies)
* Control Arm and Exploratory Arm:

  * No available data for diagnosis of cancer up to 365 days after or on the baseline visit
  * A histopathological or clinically indicated diagnosis of cancer within 365 days from the baseline visit, according to biobank database(s), or through linkage with cancer registry(ies)

Sub-Study 2

Inclusion Criteria

* At the baseline visit, 35 - 80 years old, any gender
* Not receiving treatment for or under surveillance for cancer at the baseline visit
* No indications of being monitored for or under consideration for suspected cancer at the baseline visit
* No diagnosis of cancer before or on the baseline visit or if any previous diagnosis of cancer, then cancer must have been curatively treated ≥ 5 years before the baseline visit
* At the baseline visit, available biospecimens for both EDTA-plasma and urine

Exclusion Criteria

* No available data for diagnosis of cancer up to 365 days after the baseline visit
* A subject with only a self-reported diagnosis of cancer in the 365 days after the baseline visit and absence of a histopathological or clinically indicated diagnosis of cancer, according to biobank database(s), or through linkage with cancer registry(ies)
* Subjects not meeting the specifications for the target population eventually changed during test development in Sub-Study 1. Note that these specifications are pre-specified in the Statistical Analysis Plan and will be applied if they meet pre-specified acceptance criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults between 35 to 80 years old asymptomatic for cancer and with no recent history of cancer.
Sampling Method: Probability Sample
Enrollment: 9170 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of the combined free GAGome MCED test | Within 365 days after the baseline visit
  Indicative of any-type cancer vs. no cancer diagnosis

SECONDARY OUTCOMES:
Sensitivity and specificity of the plasma free GAGome MCED test | Within 365 days after the baseline visit
  Indicative of any-type cancer vs. no cancer diagnosis
Sensitivity and specificity of the urine free GAGome MCED test | Within 365 days after the baseline visit
  Indicative of any-type cancer vs. no cancer diagnosis
Accuracy to the "putative cancer location" (PCL) model in the case (cancer) arm | Within 365 days after the baseline visit
  Accuracy to the "putative cancer location" (PCL) model in the case (cancer) arm
Overall survival (OS) in the case (cancer) arm | From baseline visit until the date of death from any cause, assessed up to 15 years
  Overall survival (OS) in the case (cancer) arm

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Gatto, PhD, Principal Investigator — Elypta AB
Locations (1):
- Elypta AB, Stockholm, Sweden